CLINICAL TRIAL: NCT05737836
Title: An Evaluation of Clinical Study Experiences of Patients With Ulcerative Colitis
Brief Title: Analyzing the Factors in Ulcerative Colitis Patients' Clinical Trial Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80979547
Record Dates: First submitted 2023-02-04; First posted 2023-02-21 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in clinical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of Ulcerative Colitis patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future Ulcerative Colitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of Ulcerative Colitis
* Ability to understand the study procedures, benefits and risks, and sign a written informed consent document.

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Women who are pregnant, intend to become pregnant, or are lactating
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ulcerative Colitis patients who are actively considering involvement in a clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to join in an Ulcerative Colitis clinical trial | 3 months
Number of Ulcerative Colitis patients who remain in clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hindryckx P, Baert F, Hart A, Magro F, Armuzzi A, Peyrin-Biroulet L; Clinical Trial Committee Clincom of the European Crohn's and Colitis Organisation (ECCO). Clinical trials in ulcerative colitis: a historical perspective. J Crohns Colitis. 2015 Jul;9(7):580-8. doi: 10.1093/ecco-jcc/jjv074. Epub 2015 Apr 25. PMID 25913641
- [Background] Sebastian S, Walker GJ, Kennedy NA, Conley TE, Patel KV, Subramanian S, Kent AJ, Segal JP, Brookes MJ, Bhala N, Gonzalez HA, Hicks LC, Mehta SJ, Lamb CA; PROTECT-ASUC Study Group. Assessment, endoscopy, and treatment in patients with acute severe ulcerative colitis during the COVID-19 pandemic (PROTECT-ASUC): a multicentre, observational, case-control study. Lancet Gastroenterol Hepatol. 2021 Apr;6(4):271-281. doi: 10.1016/S2468-1253(21)00016-9. Epub 2021 Feb 2. PMID 33545083
- [Background] Feuerstein JD, Cheifetz AS. Ulcerative colitis: epidemiology, diagnosis, and management. Mayo Clin Proc. 2014 Nov;89(11):1553-63. doi: 10.1016/j.mayocp.2014.07.002. Epub 2014 Sep 8. PMID 25199861

DOCUMENTS (1):
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT05737836/ICF_000.pdf